CLINICAL TRIAL: NCT01538459
Title: Plasma Glucose Levels With Dexamethasone as Adjuvant to Interscalene Block
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Lifespan (Other)
Collaborators: United States Naval Medical Center, Portsmouth (U.S. Federal Agency)
Responsible Party: Principal Investigator, Geoffrey Wilson, M.D., Staff Anesthesiologist, Principal Investigator, United States Naval Medical Center, Portsmouth
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NHCNE.2012.0001
Record Dates: First submitted 2012-02-20; First posted 2012-02-24 (Estimated); Last update posted 2013-05-20 (Estimated); Status verified 2013-05

CONDITIONS: Shoulder Pain; Injury of Shoulder Region; Disorder of Shoulder; Disorder of Rotator Cuff; Disorder of Tendon of Biceps
Keywords: Blood Glucose; Bupivacaine; Interscalene Nerve Block; Regional Anesthesia; Pain Blockade; Arthroscopic Surgery; Arthroscopic rotator cuff repair; Dexamethasone; Anti-Inflammatory Agents; Therapeutic Uses; Physiological Effects of Drugs; Glucocorticoids; Anesthetics, Local; Anesthetics; Sensory System Agents; Adjuvants, Anesthesia; Anesthesiology; Injections; Adult; Analgesia/methods; Brachial Plexus/drug effects; Brachial Plexus/surgery; Brachial Plexus/ultrasonography; Bupivacaine/administration & dosage; Dexamethasone/administration & dosage; Drug Therapy, Combination; Female; Humans; Male; Nerve Block/methods; Pain, Postoperative/etiology; Pain, Postoperative/prevention & control; Prospective Studies; Time Factors
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Agnosia; Pain | interventions — Dexamethasone; Calcium Dobesilate; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine (Active Comparator): 50 randomized participants in group receive 20cc 0.25% bupivacaine injected perineurally for interscalene nerve block.
  Interventions: Drug: Bupivacaine
- Dexamethasone and Bupivacaine (Experimental): 50 randomized participants in group will 8 mg(2cc of 4mg/cc solution) Dexamethasone added to 20 cc 0.25% bupivacaine in one syringe resulting in 364 µgm/cc for injection. Injected perineurally for interscalene nerve block pre-operatively.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Dexamethasone — 8mg (2cc 4mg/cc Solution) mixed with 20 cc 0.25% bupivacaine in one syringe resulting in 364 µgm/cc for injection in perineural space. One time dose during nerve block preoperatively.
  Other Names: Decadron
  Arms: Dexamethasone and Bupivacaine
Drug: Bupivacaine — Control Group receives 20 cc 0.25% bupivacaine without any adjuvants
  Arms: Bupivacaine

SUMMARY:
The purpose of this study is to determine the Finger Blood Glucose (sugar) when dexamethasone is added to a local anesthetic for a shoulder nerve block procedure. The investigators hypothesize that there is no increase in plasma glucose when 8 mg of dexamethasone is used as an adjuvant with local anesthetic to interscalene regional anesthesia. By performing finger stick blood glucose measures pre/peri and post operatively the investigators will be able to determine if any such increase exists.

DETAILED DESCRIPTION:
Patients receiving regional anesthesia for orthopedic surgeries are provided with significant pain relief in the post-operative period. Dexamethasone as an adjuvant to local anesthetic has been shown to provide increased duration of block without adverse effects. Use of steroids as adjuvants are restricted to non-diabetics due to concern for increased plasma glucose from systemic absorption. The investigators hypothesize that there will be no difference(increase) from patient baseline(preoperative plasma glucose) in plasma glucose levels up to 4 hours post nerve block in patients who receive 8 mg of dexamethasone used as an adjuvant with local anesthetic to interscalene regional anesthesia. Research has demonstrated the safety and efficacy of dexamethasone as an adjuvant to local anesthetic in peripheral nerve block. Currently there are no studies which document any plasma glucose effects(or lack of effects) from dexamethasone used as an adjuvant to regional anesthesia. Currently dexamethasone is used clinically off label by anesthesiologists as an adjuvant in association with local anesthetic for nerve block anesthesia. Once studies are completed, the investigators hope to allow diabetics to also receive the prolongation of pain relief associated with the use of steroid as an adjuvant. In addition, the increased educational and pharmacological data gleamed from the data can potentially be utilized for future studies with dexamethasone utilized perineurally.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1 or ASA 2 male or female non pregnant patients undergoing elective shoulder arthroscopy for surgical repair.

Exclusion Criteria:

* severe lung disease
* contralateral diaphragmatic paralysis
* coagulopathy
* pregnancy
* pre-existing neuropathy involving the surgical limb
* systemic use of corticosteroids for 2 weeks or longer within 6 months of surgery
* chronic opioid use (30 mg oral oxycodone equivalent per day)
* diabetes I or II
* diagnosis of "pre-diabetes"
* currently prescribed any of the oral glucose medications :sulfonylureas, meglitinides, biguanides, thiazolidinediones, alpha-glucosidase inhibitors, or DPP-4 inhibitors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2013-11 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Increased Blood Sugar after Dexamethasone added to local anesthetic for interscalene nerve block. | 4 hours
  Normal fasting blood glucose is defined by investigators as less than 100mg/dL.(current literature suggests normal is 70-100 so investigators have chosen to utilize high normal.) Any increase greater than 10%(or 10mg/dL ) would be considered a response to the dexamethasone.

SECONDARY OUTCOMES:
Pain post-operative(immediately)- both at rest and with movement(VAS Scale) | 4 hours
  Investigators will document patient pain in post-anesthesia care unit (both at rest and with movement)utilizing the VAS scale.
Time until first narcotic usage post operatively | 14 days
  Patients will be called for follow-up days 1, 2 and 14 and provided with a pain diary to document first narcotic usage.
Block Quality and Duration(time until first motor return) | 14 Days
  Patients will be called for follow up on days 1, 2 and 14 and provided with a pain diary to document the quality and duration of the motor block.
Block Quality and Duration(time until first sensory return) | 14 Days
  Patients will be called for follow up on days 1, 2 and 14 and provided with a pain diary to document the quality and duration of the sensory block.

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey W Wilson, M.D., Principal Investigator — United States Navy; Raul Masing, M.D., Principal Investigator — Lifespan
Locations (1):
- Newport Hospital, Newport, Rhode Island, United States

REFERENCES:
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Background] Thornton PC, Grant SA, Breslin DS. Adjuncts to local anesthetics in peripheral nerve blockade. Int Anesthesiol Clin. 2010 Fall;48(4):59-70. doi: 10.1097/AIA.0b013e3181f89af1. No abstract available. PMID 20881527
- [Background] Bigat Z, Boztug N, Hadimioglu N, Cete N, Coskunfirat N, Ertok E. Does dexamethasone improve the quality of intravenous regional anesthesia and analgesia? A randomized, controlled clinical study. Anesth Analg. 2006 Feb;102(2):605-9. doi: 10.1213/01.ane.0000194944.54073.dd. PMID 16428570
- [Background] Kopacz DJ, Lacouture PG, Wu D, Nandy P, Swanton R, Landau C. The dose response and effects of dexamethasone on bupivacaine microcapsules for intercostal blockade (T9 to T11) in healthy volunteers. Anesth Analg. 2003 Feb;96(2):576-82, table of contents. doi: 10.1097/00000539-200302000-00050. PMID 12538215
- [Background] Kopacz DJ, Bernards CM, Allen HW, Landau C, Nandy P, Wu D, Lacouture PG. A model to evaluate the pharmacokinetic and pharmacodynamic variables of extended-release products using in vivo tissue microdialysis in humans: bupivacaine-loaded microcapsules. Anesth Analg. 2003 Jul;97(1):124-31, table of contents. doi: 10.1213/01.ane.0000067531.49000.c1. PMID 12818954
- [Background] Drager C, Benziger D, Gao F, Berde CB. Prolonged intercostal nerve blockade in sheep using controlled-release of bupivacaine and dexamethasone from polymer microspheres. Anesthesiology. 1998 Oct;89(4):969-79. doi: 10.1097/00000542-199810000-00022. PMID 9778015
- [Background] Movafegh A, Razazian M, Hajimaohamadi F, Meysamie A. Dexamethasone added to lidocaine prolongs axillary brachial plexus blockade. Anesth Analg. 2006 Jan;102(1):263-7. doi: 10.1213/01.ane.0000189055.06729.0a. PMID 16368840
- [Background] Manchikanti L, Boswell MV, Datta S, Fellows B, Abdi S, Singh V, Benyamin RM, Falco FJ, Helm S, Hayek SM, Smith HS; ASIPP. Comprehensive review of therapeutic interventions in managing chronic spinal pain. Pain Physician. 2009 Jul-Aug;12(4):E123-98. PMID 19668281
- [Background] Holte K, Werner MU, Lacouture PG, Kehlet H. Dexamethasone prolongs local analgesia after subcutaneous infiltration of bupivacaine microcapsules in human volunteers. Anesthesiology. 2002 Jun;96(6):1331-5. doi: 10.1097/00000542-200206000-00011. PMID 12170044
- [Background] Parrington SJ, O'Donnell D, Chan VW, Brown-Shreves D, Subramanyam R, Qu M, Brull R. Dexamethasone added to mepivacaine prolongs the duration of analgesia after supraclavicular brachial plexus blockade. Reg Anesth Pain Med. 2010 Sep-Oct;35(5):422-6. doi: 10.1097/AAP.0b013e3181e85eb9. PMID 20814282
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Raj's Practical Management of Pain, 4th ed. Benzon HT, Rathmel JP, Wu CL, Turk DC, Argoff CE, eds. Philadelphia: Mosby/Elsevier, 2008.